CLINICAL TRIAL: NCT00037518
Title: An Assessment of the Calcimimetic Agent AMG 073 for the Treatment of Subjects With Parathyroid Carcinoma or Intractable Primary Hyperparathyroidism.
Brief Title: A Study of an Investigational Medication for Severe Primary Hyperparathyroidism or Parathyroid Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20000204
Record Dates: First submitted 2002-05-17; First posted 2002-05-20 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Hyperparathyroidism; Parathyroid Neoplasms
Keywords: Severe primary hyperparathyroidism; Parathyroid carcinoma
MeSH Terms: conditions — Hyperparathyroidism; Parathyroid Neoplasms; Hyperparathyroidism, Primary | interventions — Cinacalcet

INTERVENTIONS:
Drug: AMG 073

SUMMARY:
This study will assess an investigational medication for patients with severe primary hyperparathyroidism or parathyroid cancer.

ELIGIBILITY:
* Patients must have parathyroid carcinoma or severe primary hyperparathyroidism; * Abnormally elevated calcium levels above 12.5 mg/dL; * Not be pregnant or nursing; * Not have had any type of cancer other than parathyroid carcinoma within the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46
Dates: Start 2001-04

PRIMARY OUTCOMES:
Changes in serum calcium and PTH

SECONDARY OUTCOMES:
Safety and tolerability of cinacalcet

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Silverberg SJ, Rubin MR, Faiman C, Peacock M, Shoback DM, Smallridge RC, Schwanauer LE, Olson KA, Klassen P, Bilezikian JP. Cinacalcet hydrochloride reduces the serum calcium concentration in inoperable parathyroid carcinoma. J Clin Endocrinol Metab. 2007 Oct;92(10):3803-8. doi: 10.1210/jc.2007-0585. Epub 2007 Jul 31. PMID 17666472
- [Result] Marcocci C, Chanson P, Shoback D, Bilezikian J, Fernandez-Cruz L, Orgiazzi J, Henzen C, Cheng S, Sterling LR, Lu J, Peacock M. Cinacalcet reduces serum calcium concentrations in patients with intractable primary hyperparathyroidism. J Clin Endocrinol Metab. 2009 Aug;94(8):2766-72. doi: 10.1210/jc.2008-2640. Epub 2009 May 26. PMID 19470620
- [Derived] Peacock M, Bilezikian JP, Bolognese MA, Borofsky M, Scumpia S, Sterling LR, Cheng S, Shoback D. Cinacalcet HCl reduces hypercalcemia in primary hyperparathyroidism across a wide spectrum of disease severity. J Clin Endocrinol Metab. 2011 Jan;96(1):E9-18. doi: 10.1210/jc.2010-1221. Epub 2010 Oct 13. PMID 20943783
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com